CLINICAL TRIAL: NCT02327117
Title: Low Dose Peri- Operative Intra Venous Teranexamic Acid Reduces Blood Loss After Total Knee Arthroplasty: A Double Blind Randomized Placebo Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amin Nemati, Orthopedic surgery resident,Orthopedic department,Alzahra hospital,Isfahan University of Medical Sciences,Isfahan,Iran, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 392114
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Knee Arthroplasty, Total
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

ARMS (2):
- Tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic Acid
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic acid
Drug: Normal saline
  Arms: Normal Saline

SUMMARY:
Total Knee Arthroplasty (TKA) is a common orthopedic surgery usually leads to Bleeding. The null hypothesis of this study was that TA has no effect on post surgical bleeding in patients undergoes TKA.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with osteoarthritis who indicated for primary TKA.

Exclusion Criteria:

* Previous history of ceberovascular diseases
* Previous history of myocardial infarction
* Candidates for bilateral TKA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Amin Nemati, Isfahan, Isfahan, Iran

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid: Tranexamic Acid
- Normal Saline: Normal saline
Period: Overall Study
Arm/Group | Tranexamic Acid | Normal Saline
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Normal Saline | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: year] | 67.04 (8.01) | 65.66 (4.97) | 66.35 (6.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Hb Level 48 Hours After Total Knee Arthroplasty
Time Frame: 48 hours after TKA
Measure: Mean (Standard Deviation); unit: gr/dL
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 45 | 45
gr/dL | 10.92 (0.07) | 10.23 (0.98)

ADVERSE EVENTS:
Arm/Group | Tranexamic Acid | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No